CLINICAL TRIAL: NCT00664326
Title: A Phase II Uncontrolled Study of BAY73-4506 in Previously Untreated Patients With Metastatic or Unresectable Renal Cell Cancer (RCC)
Brief Title: A Phase II Uncontrolled Study of BAY73-4506 in Previously Untreated Patients With Metastatic or Unresectable RCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11726; 2008-000107-28 (EudraCT Number)
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Results first posted 2012-11-28 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib (Stivarga, BAY73-4506) (Experimental): Participants received Regorafenib 160 mg per os (po) every day (qd) for 3 weeks on 1 week off of every 4 week cycle
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Patients will be treated with BAY73-4506 160 mg po qd for 3 weeks of every 4 week cycle (i.e., 3 weeks on, 1 week off). Patients will continue treatment with BAY73-4506 until disease progression, intolerable toxicity, or patient refusal to continue with the study or investigator decision to remove the patient from study.

SUMMARY:
This is a uncontrolled, open-label, non-randomized Phase II study of oral BAY73-4506 to evaluate the response rate of BAY73-4506 in previously untreated patients with metastatic or unresectable renal cell cancer (RCC).

DETAILED DESCRIPTION:
The final analysis of efficacy will be performed after last patient has been treated for at least 6 months. Additional periodic safety and efficacy data reviews will be performed for any patients continuing to receive study drug afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >/= 18 years of age.
* Patients, who suffer from unresectable and/or metastatic, measurable predominantly clear cell RCC (renal cell carcinoma histologically) or cytologically documented.
* Patients must be previously untreated for advanced disease. Prior palliative radiation therapy is allowed if the target lesion(s) are not included within the radiation field and no more than 30% of the bone marrow is irradiated.
* Patients who have at least one uni-dimensional measurable lesion by computed tomography (CT-scan) or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST).
* Patients with "Intermediate" or "Low" risk per the Motzer score.
* Patients who have an Eastern Co-operative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate bone marrow, renal and hepatic function as assessed by the following laboratory requirements to be conducted within 7 days prior to study drug treatment

Exclusion Criteria:

* Patients who have received prior systemic treatment regimens for RCC.
* Uncontrolled/unstable cardiac disease
* Uncontrolled hypertension
* Active clinically serious infections (> Common Terminology Criteria for Adverse Events [CTCAE] grade 2 )
* History of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
* Known history or symptomatic metastatic brain or meningeal tumours
* Patients with seizure disorder requiring medication
* Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event >/= CTCAE Grade 3 within 4 weeks of first dose of study.
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-04-30 (Actual); Primary Completion 2009-05-31 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- United States (2):
  - Los Angeles, California
  - Houston, Texas
- Finland (2):
  - Helsinki
  - Turku
- France (2):
  - Nantes
  - Paris
- Germany (4):
  - Frankfurt am Main, Hesse
  - Dresden, Saxony
  - Berlin
  - Hamburg
- Poland (3):
  - Bialystok
  - Lublin
  - Poznan
- United Kingdom (5):
  - Leicester, Leicestershire
  - Bristol
  - Cambridge
  - London
  - Northwood

REFERENCES:
- [Result] Eisen T, Joensuu H, Nathan PD, Harper PG, Wojtukiewicz MZ, Nicholson S, Bahl A, Tomczak P, Pyrhonen S, Fife K, Bono P, Boxall J, Wagner A, Jeffers M, Lin T, Quinn DI. Regorafenib for patients with previously untreated metastatic or unresectable renal-cell carcinoma: a single-group phase 2 trial. Lancet Oncol. 2012 Oct;13(10):1055-62. doi: 10.1016/S1470-2045(12)70364-9. Epub 2012 Sep 6. PMID 22959186
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female untreated participants, who were at least 18 years of age, with metastatic and/or unresectable, measurable predominantly clear cell renal cell cancer (RCC) histologically or cytologically documented could participate in this study at 18 centers in 6 countries.
Pre-assignment Details: Of 64 enrolled participants, 49 received study medication, and 15 were screen failures due to protocol violation (12 participants), withdrawal of consent (1 participant), adverse event (2 participants).
Period: Overall Study
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Started | 49
Completed | 1 (transitioned to rollover study)
Not Completed | 48
Not completed — Adverse Event | 14
Not completed — Noncompliance with study medication | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Other Reasons | 3
Not completed — Death | 2
Not completed — Disease Progression/Recurrence/Relapse | 24

BASELINE CHARACTERISTICS:
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: Years] | 62.0 [40 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 27
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — The ECOG PS ranged from Grades 0 to 5 (death). Grade 0 (fully active, able to carry on all pre-diseases performance without restriction) and Grade 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature) were inclusion criteria.
  Participants
    0 | 30
    1 | 19
Overall Motzer Score [Count of Participants; unit: Participants] — The Motzer score (high/poor risk, intermediate risk, low risk) is based on the number of the following poor prognostic features a participant possessed: ECOG >2, serum lactate dehydrogenase concentration > 1.5 times the upper limit of normal, hemoglobin < lower limit of normal, corrected calcium concentration > 10 mg/dl, and absence of prior nephrectomy. Participants who had none of these features = low risk; participants with 1 or 2 of these features = intermediate risk; participants with 3 or more of these features = high/poor risk and were excluded from participating in the study.
  Participants
    Low | 24
    Intermediate | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: Objective tumor response of a participant was defined as the best tumor response (confirmed Complete Response [CR, tumor disappears] or Partial Response [PR, sum of lesion sizes decreased at least 30% from baseline]) observed during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) committee.
Time Frame: From start of treatment of the first participant until database cut-off approximately 13 months later (13May2008 - 31May2009). Assessed every 8 weeks for 6 months, then every 12 weeks
Population: Evaluable for response (Primary analysis population)
Measure: Number; unit: Percentage of participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 48
Percentage of participants | 31.3

2. Primary Outcome: Tumor Response
Description: Tumor response of a participant was defined as the best tumor response (confirmed Complete Response [CR, tumor disappears], Partial Response [PR, sum of lesion sizes decreased at least 30% from baseline], Stable Disease [SD, steady state of disease], or Progressive Disease [PD, sum of lesion sizes increased at least 20% from smallest sum on study or new lesions]) observed during trial period assessed according to the RECIST committee.
Time Frame: as for outcome 1
Population: Evaluable for response (Primary analysis population)
Measure: Number; unit: Percentage of participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 48
Percentage of participants
  Complete Response (CR) | 0.0
  Partial Response (PR) | 31.3
  Stable Disease (SD) | 50.0
  Progressive Disease (PD) | 10.4
  Not Assessable | 8.3

3. Secondary Outcome: Disease Control
Description: Disease control was defined as the percentage of participants who had a best response rating of CR (tumor disappears), PR (sum of lesion sizes decreased at least 30% from baseline), or SD (steady state of disease) that was maintained for at least 28 days from the first demonstration of that rating.
Time Frame: as for outcome 1
Population: Evaluable for response (Primary analysis population)
Measure: Number; unit: Percentage of participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 48
Percentage of participants | 62.5

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was calculated as the time from the first date of receiving study medication to death, due to any cause. Participants alive at the time of analysis were censored at their last date of follow-up.
Time Frame: From start of treatment of the first participant until database cut-off approximately 13 months later (13May2008 - 31May2009).
Population: intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 49
Days | NA [285 to NA] — Not estimable due to censored data.

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was calculated as time from first date of receiving study drug until date of first observed disease progression (PD) (radiological or clinical, whichever was earlier) or death due to any cause, if death occurred before PD was documented. The actual date of tumor assessments (i.e., date on which radiological procedure was performed, rather than scheduled date) was used for this calculation to determine both the event date and censoring date. Patients without PD or death at time of analysis were censored at last date of tumor evaluation.
Time Frame: as for outcome 1
Population: intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 49
Days | 251 [160 to NA] — Not estimable due to censored data.

6. Secondary Outcome: Time to Progression (TTP)
Description: TTP was calculated as time from first date of receiving study drug until date of first documented disease progression (PD) (radiological or clinical, whichever was earlier). The actual date of tumor assessments (i.e., date on which radiological procedure was performed, rather than the scheduled date) was used for this calculation to determine both the event date and censoring date. Patients without PD at time of analysis were censored at last date of tumor evaluation.
Time Frame: as for outcome 1
Population: intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 49
Days | 251 [167 to NA] — Not estimable due to censored data.

7. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the first documented objective response of PR or CR, whichever was earlier, to disease progression or death (if death occurred before progression was documented). Duration of response for subjects who had not progressed or died at the time of analysis were censored at the date of their last tumor assessment.
Time Frame: as for outcome 1
Population: Only subjects from ITT population with a response of CR or PR were included in this evaluation.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 15
Days | NA [140 to NA] — Not estimable due to censored data.

8. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of SD was calculated as the time from the first date of receiving study drug until the date of documented PD or the last observation if the subject did not progress. Subjects without disease progression at the time of analysis were censored at the last date of tumor evaluation.
Time Frame: as for outcome 1
Population: Subjects from ITT population who achieved objective response of CR or PR were excluded from this evaluation.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 29
Days | 172 [107 to NA] — Not estimable due to censored data.

9. Other Pre Specified Outcome: Objective Tumor Response (Update)
Description: Objective tumor response of a participant was defined as the best tumor response (confirmed Complete Response [CR, tumor disappears] or Partial Response [PR, sum of lesion sizes decreased at least 30% from baseline]) observed during trial period assessed according to the RECIST committee.
Time Frame: From start of treatment of the first participant until database cut-off approximately 37 months later (13May2008 - 1Jun2011). Assessed every 8 weeks for 6 months, then every 12 weeks
Population: Evaluable for response (Primary analysis population)
Measure: Number; unit: Percentage of participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 48
Percentage of participants | 39.6

10. Other Pre Specified Outcome: Tumor Response (Update)
Description: as for outcome 2
Time Frame: as for outcome 9
Population: Evaluable for response (Primary analysis population)
Measure: Number; unit: Percentage of participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 48
Percentage of participants
  Complete Response (CR) | 0.0
  Partial Response (PR) | 39.6
  Stable Disease (SD) | 41.7
  Progressive Disease (PD) | 10.4
  Not Assessable | 8.3

11. Other Pre Specified Outcome: Disease Control (Update)
Description: as for outcome 3
Time Frame: as for outcome 9
Population: Evaluable for response (Primary analysis population)
Measure: Number; unit: Percentage of participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 48
Percentage of participants | 62.5

12. Other Pre Specified Outcome: Overall Survival (Update)
Description: as for outcome 4
Time Frame: From start of treatment of the first participant until database cut-off approximately 37 months later (13May2008 - 1Jun2011).
Population: intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 49
Days | NA [735 to NA] — Not estimable due to censored data.

13. Other Pre Specified Outcome: Progression-free Survival (Update)
Description: as for outcome 5
Time Frame: as for outcome 9
Population: intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 49
Days | 335 [167 to 438]

14. Other Pre Specified Outcome: Time to Progression (Update)
Description: as for outcome 6
Time Frame: as for outcome 9
Population: intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 49
Days | 335 [167 to 454]

15. Other Pre Specified Outcome: Duration of Response (Update)
Description: as for outcome 7
Time Frame: as for outcome 9
Population: Only subjects from ITT population with a response of CR or PR were included in this evaluation.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 19
Days | 428 [250 to 540]

16. Other Pre Specified Outcome: Duration of Stable Disease (Update)
Description: as for outcome 8
Time Frame: as for outcome 9
Population: Subjects from ITT population who achieved objective response of CR or PR were excluded from this evaluation.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)
Number analyzed (Participants) | 25
Days | 119 [105 to 335]

ADVERSE EVENTS:
Description: Acronyms used in Adverse events section: Gastrointestinal (GI), Not Otherwise Specified (NOS), Absolute Neutrophil Count (ANC), Common Terminology Criteria for Adverse Events (CTCAE).
Groups:
- Regorafenib (BAY73-4506): Subjects received regorafenib 160 mg po qd for 3 weeks of every 4 week cycle (3 weeks on, 1 week off).
Arm/Group | Regorafenib (BAY73-4506)
All-Cause Mortality (participants affected / at risk) | 39/49
Serious Adverse Events (participants affected / at risk) | 32/49
Other Adverse Events (participants affected / at risk) | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (BAY73-4506) (N=49)
Angina unstable (Cardiac disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (3)
Renal failure (Renal and urinary disorders) | 4 (7)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Tumour excision (Surgical and medical procedures) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (BAY73-4506) (N=49)
Anaemia (Blood and lymphatic system disorders) | 5 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (11)
Abdominal pain (Gastrointestinal disorders) | 13 (37)
Abdominal pain upper (Gastrointestinal disorders) | 8 (28)
Constipation (Gastrointestinal disorders) | 17 (112)
Diarrhoea (Gastrointestinal disorders) | 24 (215)
Dyspepsia (Gastrointestinal disorders) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 4 (5)
Glossodynia (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 16 (46)
Oral pain (Gastrointestinal disorders) | 6 (35)
Stomatitis (Gastrointestinal disorders) | 15 (108)
Vomiting (Gastrointestinal disorders) | 13 (29)
Chest pain (General disorders) | 7 (19)
Chills (General disorders) | 3 (6)
Fatigue (General disorders) | 22 (192)
Mucosal inflammation (General disorders) | 6 (11)
Oedema peripheral (General disorders) | 4 (13)
Pain (General disorders) | 6 (31)
Pyrexia (General disorders) | 9 (14)
Bronchitis (Infections and infestations) | 3 (3)
Infection (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 9 (21)
Oral candidiasis (Infections and infestations) | 3 (7)
Rhinitis (Infections and infestations) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 4 (6)
Urinary tract infection (Infections and infestations) | 6 (13)
Amylase increased (Investigations) | 4 (12)
Blood creatinine increased (Investigations) | 3 (7)
Lipase increased (Investigations) | 7 (29)
Weight decreased (Investigations) | 8 (86)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (13)
Decreased appetite (Metabolism and nutrition disorders) | 16 (104)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (120)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (55)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (25)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (53)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (23)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (85)
Ageusia (Nervous system disorders) | 3 (4)
Dizziness (Nervous system disorders) | 4 (7)
Dysgeusia (Nervous system disorders) | 4 (14)
Headache (Nervous system disorders) | 14 (47)
Neuropathy peripheral (Nervous system disorders) | 4 (8)
Paraesthesia (Nervous system disorders) | 4 (61)
Insomnia (Psychiatric disorders) | 6 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (15)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 (50)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (48)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (139)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (77)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (19)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (8)
Palmar erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 34 (402)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (16)
Rash (Skin and subcutaneous tissue disorders) | 17 (74)
Rash generalised (Skin and subcutaneous tissue disorders) | 3 (4)
Hypertension (Vascular disorders) | 25 (338)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12-18 months after database lock at the earliest. Bayer will have 30-45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable).

No publication of single center data should be done prior of publication if multi-center data.